CLINICAL TRIAL: NCT04649814
Title: Finnish Spinal Cord Injury Study (FinSCI)
Acronym: FinSCI
Status: Completed | Type: Observational
Sponsor: The Finnish Association of People with Physical Disabilities (Other)
Collaborators: Helsinki University Central Hospital (Other); Tampere University Hospital (Other); Oulu University Hospital (Other); The Finnish Association of Spinal Cord Injured Akson (Unknown); Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Sponsor
Other Study IDs: 42106
Record Dates: First submitted 2018-08-30; First posted 2020-12-02 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Spinal Cord Injuries; Health, Subjective
Keywords: patient reported outcomes; ICF; Survey; Interview
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Questionnaire for all, interview for part of the respondents.
  Other Names: interview

SUMMARY:
The purpose of the Finnish Spinal Cord Injury Study (FinSCI) is to identify factors related to the health and functioning of people with spinal cord injury (SCI), their challenges with accessibility and how such factors are interconnected. The International Classification of Functioning, Disability and Health (ICF) is used in the study as a structured framework. The study participants will be recruited from three SCI outpatient clinics, which together are responsible for the life-time care of the SCI population in Finland.

Mixed methods are used including a questionnaire and interviews. The survey will be formed from patient-reported instruments; SCI-specified Spinal Cord Injury Secondary Condition Scale, Spinal Cord Independence Measure, Nottwil Environmental Factors Inventory Short Form and selected items of the generic instruments of Patient-Reported Outcomes Measurement Information System and National study of health, well-being and service. The survey covers 51 ICF categories. The study results can help develop care and rehabilitation policies with SCI, the planning of training models and information provided to various parties involved.

DETAILED DESCRIPTION:
The detailed description of the protocol has been published. Please, see the reference Tallqvist et al.

ELIGIBILITY:
Inclusion Criteria:

* 16 years or over
* Traumatic or non-traumatic SCI
* ASIA-classification A,B,C tai D
* Time since onset of SCI over 6 months
* Client of HUS, Tays or Oys SCI outpatient clinic

Exclusion Criteria:

* Innate SCI
* Progressive new non-traumatic SCI
* Neurodegenerative disease
* Multiple sclerosis amyotrophic lateral sclerosisGuillain-Barre syndrome Institutional care

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Acute care, immediate rehabilitation and life-long multi-professional follow-up, care and rehabilitation of SCI have been centralised at 3 university hospitals: Oulu (OYS), Tampere (Tays) and Helsinki (HUS) university hospitals. They serve the whole SCI-population, both previously and newly injured, in their hospital district areas. The study participants were selected by exploring the patient registries in OYS, Tays and HUS. A more systematic data collection of the SCI population started in different outpatient clinics at different times (Tays 5/2011, OYS 1/2012 and in HUS 8/2013). The selection of patients for the study performed from the start of the systematic data collection and lasted in Tays and OYS till the end of 2017, and in HUS - till the end of June 2018.
Sampling Method: Non-Probability Sample
Enrollment: 1773 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Cohort Survey of Health, Functioning, and accessibility of spinal cord injury population in Finland | 1.2.-31.7.2019
  Survey includes parameters of secondary conditions of spinal cord injury, independency, environmental factors, health, well-being and services

CONTACTS AND LOCATIONS:
Overall Officials: Hiekkala, PhD, Study Director — Research Director
Locations (1):
- The Finnish Association of People with Physical Disabilities, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: Yes
We share study protocol.
Supporting Information: Study Protocol
Time Frame: The protocol has been published.
Access Criteria: To be able to log in Internet.
URL: https://www.medicaljournals.se/jrm/content/abstract/10.2340/16501977-2539

REFERENCES:
- [Background] Tallqvist S, Anttila H, Kallinen M, Koskinen E, Hamalainen H, Kauppila AM, Tackman A, Vainionpaa A, Arokoski J, Hiekkala S. Health, functioning and accessibility among spinal cord injury population in Finland: Protocol for the FinSCI study. J Rehabil Med. 2019 Apr 1;51(4):273-280. doi: 10.2340/16501977-2539. PMID 30805657
- [Background] Tallqvist S, Kauppila AM, Vainionpaa A, Koskinen E, Bergman P, Anttila H, Hamalainen H, Tackman A, Kallinen M, Arokoski J, Hiekkala S. Prevalence of comorbidities and secondary health conditions among the Finnish population with spinal cord injury. Spinal Cord. 2022 Jul;60(7):618-627. doi: 10.1038/s41393-021-00704-7. Epub 2021 Sep 11. PMID 34511604
- [Background] Majamaki K, Tallqvist S, Vainionpaa A, Koskinen E, Kauppila AM, Bergman P, Anttila H, Hamalainen H, Tackman A, Kallinen M, Arokoski J, Hiekkala S. Functional independence in the Finnish spinal cord injury population. Spinal Cord. 2022 Jul;60(7):628-634. doi: 10.1038/s41393-021-00700-x. Epub 2021 Sep 15. PMID 34526631
- [Background] Eskola K, Koskinen E, Anttila H, Tallqvist S, Bergman P, Kallinen M, Hamalainen H, Kauppila AM, Tackman A, Vainionpaa A, Arokoski J, Rajavaara M, Hiekkala S. Health-related factors for work participation in persons with spinal cord injury in Finland. J Rehabil Med. 2022 Feb 3;54:jrm00255. doi: 10.2340/jrm.v53.59. PMID 34888701
- [Background] Poutanen J, Anttila H, Tallqvist S, Kallinen M, Koskinen E, Hamalainen H, Kauppila AM, Tackman A, Vainionpaa A, Arokoski J, Hiekkala S. Physical health among the Finnish spinal cord injury population according to the Patient Reported Outcome Measurement Information System (PROMIS(R)). J Spinal Cord Med. 2022 Nov;45(6):865-873. doi: 10.1080/10790268.2021.1989184. Epub 2021 Nov 2. PMID 34726579
- See also: Project webpage — https://www.invalidiliitto.fi/finsci-selkaydinvammaisten-henkiloiden-terveys-ja-toimintakyky-seka-haasteet-esteettomyydessa